CLINICAL TRIAL: NCT00176826
Title: In-vivo T-cell Depletion and Hematopoietic Stem Cell Transplantation for Life-Threatening Immune Deficiencies and Histiocytic Disorders
Brief Title: T-Cell Depletion and Stem Cell Transplant for Immune Deficiencies and Histiocytic Disorders
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Replaced by another protocol
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMN-MT2000-21; 0010M66781 (Other: Institutional Review Board, University of Minnesota); NCT00973843 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2015-05

CONDITIONS: Hemophagocytic Lymphohistiocytosis; X-Linked Lymphoproliferative Disorders; Chediak-Higashi Syndrome; Griscelli Syndrome; Immunologic Diseases; Langerhans-Cell Histiocytosis; Hematologic Diseases
Keywords: Stem Cell Transplant; T-cell depletion; immune deficiencies; Busulfan pharmacokinetics; Non-Malignant Hematological Disorders
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Lymphoproliferative Disorders; Chediak-Higashi Syndrome; Immune System Diseases; Histiocytosis, Langerhans-Cell; Hematologic Diseases | interventions — Stem Cell Transplantation; Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intent-To-Treat (Experimental): Patients who were treated with chemotherapies (myeloablative conditioning regimen) and stem cell transplant. Busulfan intravenously for 4 days followed by cyclophosphamide intravenously for 4 days. Rabbit ATG is given intravenously for 4 doses pre-transplant.
  Interventions: Procedure: Stem Cell Transplant; Drug: Myeloablative conditioning regimen

INTERVENTIONS:
Procedure: Stem Cell Transplant — Infusion of hematopoietic stem cells (bone marrow, cord blood, peripheral blood stem cells) following myeloablative conditioning regimen.
  Other Names: HSCT
Drug: Myeloablative conditioning regimen — Busulfan intravenously for 4 days followed by cyclophosphamide intravenously for 4 days. Rabbit ATG is given intravenously for 4 doses pre-transplant.
  Other Names: Busulfex; Cytoxan; ATG

SUMMARY:
The hypothesis is to determine if a preparative regimen of busulfan, cyclophosphamide, and antithymocyte globulin (ATG) plus allogeneic stem cell transplantation will be effective in the treatment of immune deficiencies and histiocytic disorders.

DETAILED DESCRIPTION:
Subjects will begin chemotherapy as a preparative regimen, which is intended to completely eliminate their defective immune system and bone marrow. The preparative regimen consists of the chemotherapy drugs (busulfan, cyclophosphamide, and antithymocyte globulin (ATG)).

Transplantation: subjects will then have a source of blood stem cells (bone marrow) from their donor administered into their catheter. Medication will be given to help prevent Graft-Versus Host Disease (GVHD). The ATG will help to deplete the donor stem cells of the type of cells that can cause GVHD and will also help to promote engraftment of the new stem cells.

Recovery Phase: The second phase of treatment consists of a period after transplantation during which we wait for the return of bone marrow function. This usually takes two to four weeks. Subjects will be given a blood cell growth factor, G-CSF, to help speed recovery of the white blood cells and potentially decrease the risk of infection and decrease the time until the bone marrow recovers.

ELIGIBILITY:
Inclusion Criteria:

* Any patient from birth to < 55 years of age fulfilling the following criteria will be eligible for this study.
* Patients meeting clinical diagnostic criteria for Hemophagocytic Lymphohistiocytosis (HLH)
* Patients meeting clinical diagnostic criteria or genetic diagnosis of X-linked lymphoproliferative disorder (XLP) and whose disease is ACTIVE but STABLE, or NON-ACTIVE/QUIESCENT.
* Patients with Chediak-Higashi Syndrome who meet the following diagnostic criteria and whose disease is ACTIVE but STABLE, or NON-ACTIVE/QUIESCENT as defined in Appendix V of the study protocol.
* Patients with Viral Associated Hemophagocytic Syndrome (VAHS) - if relapsed after other therapy or supportive care. Diagnostic criteria as above for HLH. Disease status must be ACTIVE but STABLE, or NON-ACTIVE/QUIESCENT as defined in Appendix V. It is cautioned that many patients with HLH or familial hemophagocytic lymphohistiocytosis (FHL) will have a viral infection at time of initial presentation and may therefore be misdiagnosed as having VAHS.
* Griscelli Syndrome
* Primary immune deficiencies with non-genotypic identical donors only.
* Progressive Langerhans cell histiocytosis unresponsive to standard therapy.
* Other non-malignant hematological disorders in which stem cell transplant with a myeloablative regimen is indicated.
* Diamond Blackfan Anemia if transfusion dependent
* Schwachman Diamond Syndrome: with cytopenias or transformation to myelodysplastic syndrome (MDS)
* Kostman's Syndrome (if ANC <500 without GCSF support, or transformation to MDS)
* Congenital dyserythropoietic anemia if transfusion dependent
* Amegakaryocytic thrombocytopenia if baseline platelet counts <20,000 or requiring transfusions.
* Cardiac, hepatic, renal and pulmonary function deemed adequate for high dose chemotherapy with stem cell rescue as per institutional standards. General guidelines are as follows:

  * Cardiac: Asymptomatic or, if symptomatic, then left ventricular ejection fraction at rest must be > 40% and must improve with exercise, or shortening fraction by echocardiogram must be within institutional normals
  * Hepatic: < 3 x normal SGOT and < 2.5 mg/dL serum bilirubin
  * Renal: Serum creatinine within normal range, or if serum creatinine outside normal range then creatinine clearance or glomerular filtration study should be > 50% of normal.
  * Pulmonary: Asymptomatic or, if symptomatic, diffusing capacity of the lung for carbon monoxide (DLCO) > 45% of predicted (corrected for hemoglobin). For children unable to perform pulmonary function testing, then oxygen saturation should be >95%.
* Availability of a suitable allogeneic bone marrow donor as per current institutional guidelines for non-T cell depleted hematopoietic stem cell transplant (HSCT).
* Patients who have undergone previous stem cell transplant (SCT) and failed engraftment or who had relapse of their disease are considered eligible if they meet other eligibility criteria and if the second SCT would occur 6 months or more after the first. If the first SCT preparative regimen was of a non-myeloablative intensity then the second SCT could be performed earlier when the acute toxicity from that procedure was resolved.

Exclusion Criteria:

* Patients who are moribund or whose life expectancy is severely limited by disease other than their underlying disorder. Karnofsky performance status < 70% or Lansky < 50% for patients < 16 years.
* Patients with hemophagocytic disorders secondary to underlying malignancy.
* Patients who have ACTIVE/UNSTABLE disease as defined in Appendix V.
* Significant active infections, including Human Immunodeficiency Virus (HIV).
* Age > 55 years.
* Not providing informed consent.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2000-09; Primary Completion 2012-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, MD, Principal Investigator — University of Minnesota Medical Center
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the clinic or hospital where they were being seen for their disease. The study was discussed with them at the time that treatment options were being presented.
Pre-assignment Details: Patients had to have a suitable donor identified prior to the subject starting the conditioning regimen.
Period: Overall Study
Arm/Group | Intent-To-Treat
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.7 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Time to Transplant Engraftment
Time Frame: Day 100 Post Transplant
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
days | 19.8 (5.2)

2. Secondary Outcome: Number of Patients With Treatment Related Mortality.
Time Frame: Day 100 Post Transplant
Measure: Number; unit: participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
participants | 6

3. Secondary Outcome: Number of Patients Surviving (Disease-free)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
participants | 14

4. Secondary Outcome: Number of Patients With Grade II-IV Graft-Versus-Host Disease (GVHD)
Time Frame: Day 100 Post Transplant
Measure: Number; unit: participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
participants | 4

5. Secondary Outcome: Number of Patients With Graft Failure
Time Frame: Day 100 Post transplant
Measure: Number; unit: participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
participants | 2

6. Secondary Outcome: Number of Patients With III-IV Graft-Versus-Host Disease (GVHD)
Time Frame: Day 100 Post Transplant
Measure: Number; unit: participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
participants | 1

7. Secondary Outcome: Number of Patients Surviving (Disease-free)
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
participants | 10

ADVERSE EVENTS:
Time Frame: From the time consent was signed to the end of follow-up, which was 3 years.
Arm/Group | Intent-To-Treat
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-To-Treat (N=22)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Death (General disorders) | 1 (1) — Multi-organ failure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes